CLINICAL TRIAL: NCT01649310
Title: Effects of Whole Body Vibration Training in Chronic Obstructive Pulmonary Disease (COPD) Patients: a Randomized Controlled Trial
Brief Title: Whole Body Vibration in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Patrícia Érika de Melo Marinho, Professor, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Patricia
Record Dates: First submitted 2012-06-18; First posted 2012-07-25 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Chronic obstructive pulmonary disease (COPD); Muscle strenght; Aged
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WVB Training (Experimental)
  Interventions: Other: whole body vibration

INTERVENTIONS:
Other: whole body vibration — Exercises on the platform will be made in semi-squat position, static. In the first month training will be held for 10 minutes for the exercises on the platform, 30 seconds of vibration of low intensity, interspersed with rest 60 seconds while standing beside the platform. In the second month training will be held for 15 minutes, lasting 60 seconds of vibration and 30 seconds of rest in standing beside the platform. For the first two weeks training will have low intensity and the last two weeks training will have higher vibration. In the third month, training will be held for 20 minutes, 60 seconds of vibration and 30 seconds of rest while standing beside the platform. The intensity of the vibration will be high.
  Other Names: Equipment: Power Plate my3

SUMMARY:
The whole body vibration offers better treatment adherence among the elderly, minimizing effort and additional stress to the cardiovascular system and skeletal muscles compared to conventional exercise programs.

Hypothesis: Patients with COPD undergoing a training program on the whole body vibration show better performance in the 6MWT and improvement in muscle strength.

DETAILED DESCRIPTION:
In the elderly and in COPD patients weight loss includes sarcopenia, resulting from aging itself or due to disuse or disease states associated with and represents the reduction in muscle mass, leading to decreased strength and endurance, with repercussions on the functional abilities of the same. It reduces the power and muscle strength with aging which represent decreasing to carry out daily physical tasks.

In COPD, exacerbations worsen the loss of muscle mass, affecting the respiratory and peripheral muscles, exercise capacity and survival rates, and in the case of severe malnutrition in advanced cases of the disease, the implications of this state are disability which occur between 10-15% in those with mild obstruction and 25% in moderate to severe obstructive and are associated with worse prognosis.

The whole body vibration could be an efficient combination of training methods for elderly patients and is based on the generation of sinusoidal vibrations offered by a platform, which stimulates the muscle spindles resulting in activation of neurons α engines and develop muscle contractions, presenting itself as an alternative to conventional treatment for muscular endurance as well as improving physical fitness

ELIGIBILITY:
Inclusion Criteria:

* Smoking history, occupational or environmental exposure to pollutants and / or cough, hypersecretion or dyspnea,
* FEV1 <80% predicted and postbronchodilator FEV1/FVC <70% to confirm the diagnosis of airway obstruction air not fully reversible bronchodilator therapy,
* Have the ability to perform the walk test, 6 minutes, absence of comorbidities that preclude the achievement of effort (hypertension, severe pulmonary hypertension, myocardial infarction, congestive heart failure, severe dyspnea)
* Preserved cognitive functioning,
* Clinically stable during the study period

Exclusion Criteria:

* Have cognitive impairment, hearing or visual compromise the response to the questionnaires used in this study
* Make modifications to the appliance neuro-musculo-skeletal system that prevents the completion of the 6MWT
* Be participating in physical activity programs.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2012-02; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Walked distance in 6MWT | Increase in distance walked at baseline and 3 months
  Change from baseline in distance walked test 6-minute walk test at 3 months.

SECONDARY OUTCOMES:
Respiratory muscle strength | Change from baseline in respiratory muscle strength at 3 months
  Increase in respiratory muscle strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Background] Gloeckl R, Heinzelmann I, Baeuerle S, Damm E, Schwedhelm AL, Diril M, Buhrow D, Jerrentrup A, Kenn K. Effects of whole body vibration in patients with chronic obstructive pulmonary disease--a randomized controlled trial. Respir Med. 2012 Jan;106(1):75-83. doi: 10.1016/j.rmed.2011.10.021. Epub 2011 Nov 21. PMID 22104540
- [Background] Pleguezuelos E, Perez ME, Guirao L, Samitier B, Costea M, Ortega P, Gonzalez MV, Del Carmen VA, Ovejero L, Moreno E, Miravitlles M. Effects of whole body vibration training in patients with severe chronic obstructive pulmonary disease. Respirology. 2013 Aug;18(6):1028-34. doi: 10.1111/resp.12122. PMID 23692550
- [Derived] Braz Junior DS, Dornelas de Andrade A, Teixeira AS, Cavalcanti CA, Morais AB, Marinho PE. Whole-body vibration improves functional capacity and quality of life in patients with severe chronic obstructive pulmonary disease (COPD): a pilot study. Int J Chron Obstruct Pulmon Dis. 2015 Jan 12;10:125-32. doi: 10.2147/COPD.S73751. eCollection 2015. PMID 25624756